CLINICAL TRIAL: NCT05950906
Title: A Two-Part Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetics of PDM608 in Healthy Adult Subjects
Brief Title: Study to Assess PDM608 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calibr, a division of Scripps Research (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Alzheimer's Drug Discovery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBR-PDM608-3001
Record Dates: First submitted 2023-05-22; First posted 2023-07-18 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Part 1 Cohorts 1-5 will assess single ascending doses (SAD) of subcutaneous administration PDM608. Part 2 will assess multiple ascending doses (MAD) administrations given once weekly for 4 weeks in up to 4 cohorts of participants. The parts of the study are not required to be conducted entirely sequentially, provided that this is justified by PK and safety data obtained from completed cohorts. The first MAD cohort will not start until data are available from SAD Cohort 3 and dosing for each MAD cohort will not exceed the a dose level previously deemed safe in a SAD cohort.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study; treatment assignment will not be known to the subjects, the Sponsor and staff involved in the clinical evaluation of the subjects and the analysis of data. The randomization schedule and disclosure envelopes will be generated by an unblinded statistician. The unblinded statistician will not be involved in decisions relating to populations for analysis prior to unblinding. Prior to database lock and unblinding, all original randomization materials including the original final signed and dated randomization schedule will be held by the Quality Assurance department at the study site. The Data Sciences department will not have access to the randomization schedule before database lock/unblinding. There may be instances where interim data has the potential to reveal treatment. In these cases, every effort will be made by the unblinded pharmacokinetic scientist to maintain blinding by appropriate presentation of data to the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 SAD SC PDM608 (Experimental): Single ascending dose, subcutaneous administration of PDM608
  Interventions: Drug: PDM608
- Part 1 SAD SC Placebo (Placebo Comparator): Single ascending dose, subcutaneous administration of matching placebo
  Interventions: Drug: Placebo
- Part 2 MAD SC PDM608 (Experimental): Multiple ascending dose, subcutaneous administration of PDM608 once weekly for 4 weeks.
  Interventions: Drug: PDM608
- Part 2 MAD SC Placebo (Placebo Comparator): Multiple ascending dose, subcutaneous administration of placebo once weekly for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PDM608 — PDM608 subcutaneous at single or multiple dose(s) assigned by cohort
  Arms: Part 1 SAD SC PDM608; Part 2 MAD SC PDM608
Drug: Placebo — Placebo subcutaneous at single or multiple dose(s) to match PDM608 administration.
  Arms: Part 1 SAD SC Placebo; Part 2 MAD SC Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of PDM608 in healthy adult subjects.

DETAILED DESCRIPTION:
This is a 2-part, single-center, first-in-human study of single ascending doses (SAD; Part 1) and multiple ascending doses (MAD; Part 2) of PDM608 in healthy adult subjects.

Part 1 is a double-blind, randomized, placebo-controlled assessment of subcutaneous (SC) SAD administrations of PDM608 across 5 cohorts of subjects. All SAD cohorts will follow a sentinel design. Following completion of each cohort, safety and tolerability data through 96 hours post-dose will be reviewed to determine whether to progress to the next dose level and the dose level for the next cohort.

Part 2 is a double-blind, randomized, placebo-controlled assessment of SC MAD administrations (once weekly for 4 weeks) of PDM608 across up to 4 cohorts of subjects. Following completion of each cohort the safety and tolerability data 96 hours post last dose will be reviewed to determine whether to progress to the next dose level and the dose level to be administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men, or women of non-childbearing potential
* Must agree to use an adequate method of contraception
* Body mass index (BMI) of 18.0 to 33.0 kg/m2 as measured at screening

Exclusion Criteria:

* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Significant allergy requiring treatment
* History of clinically significant autoimmune, cardiovascular, renal, hepatic, chronic respiratory or GI disease (except cholecystectomy), neurological or psychiatric disorder, illness/infection/hospitalization or surgical procedure within 30 days prior to first dose of study drug or any uncontrolled medical illness as judged by the investigator
* Have poor venous access that limits phlebotomy
* Evidence of current SARS-CoV-2 infection or exposure to confirmed infection within 10 days prior to the first dose of study drug
* Clinically significant abnormal clinical chemistry, hematology or urinalysis
* Hepatitis B, Hepatitis C, HIV, TB
* Renal impairment
* Pregnant or lactating women or men with pregnant or lactating partners
* Received any IMP in a clinical research study within 5 half-lives or within 30 days prior to first dose (whichever is longer)
* Taking any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g per day acetaminophen and HRT) in the 14 days or 5 half-lives (whichever is longer) before IMP administration
* COVID-19 vaccine within 14 days prior to first dose or have a COVID-19 vaccine scheduled between their first dose of IMP and last dose of IMP.
* Drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in men >21 units per week and women >14 units per week (1 unit = 12 oz 1 bottle/can of beer, 1 oz 40% spirit or 5 oz glass of wine)
* Positive alcohol urine test at screening or first admission
* Current and within the last six months-smokers, e-cigarettes and nicotine replacement users
* Donation of blood within 2 months or donation of plasma within 7 days prior to first dose of study medication
* Subjects who are, or are immediate family members of, a study site or Sponsor employee

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-03-17 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences-Miami, Inc, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant enrollment was reported as a combined arm (reporting PDM608 and Placebo subjects) to in sections where there is no major benefit to differentiate between treatment vs placebo. Comments were added to Part 2 MAD SC Placebo Cohort 2 to denote that the two subjects who didn't complete the study were assigned to receive active treatment. For the PK and ADA, analysis was only done on subjects who received PDM608.
Groups:
- Part 1 SAD SC PDM608 Cohort 1: One time subcutaneous administration of 350 ug of PDM608. 6 subjects received PDM608
- Part 1 SAD SC Placebo Cohort 1: One time subcutaneous administration of 350 ug of PDM608. 2 subjects received Placebo.
- Part 1 SAD SC PDM608 Cohort 2; Part 1 SAD SC Placebo Cohort 2: One time subcutaneous administration of 1050 ug of PDM608.
  2 subjects received Placebo.
- Part 1 SAD SC PDM608 Cohort 3: One time subcutaneous administration of 3150 ug of PDM608.
  6 subjects received PDM608.
- Part 1 SAD SC Placebo Cohort 3: One time subcutaneous administration of 3150 ug of PDM608.
  2 subjects received Placebo.
- Part 1 SAD SC PDM608 Cohort 4: One time subcutaneous administration of 6300 ug of PDM608.
  6 subjects received PDM608.
- Part 1 SAD SC Placebo Cohort 4: One time subcutaneous administration of 6300 ug of PDM608.
  2 subjects received Placebo.
- Part 1 SAD SC PDM608 Cohort 5: One time subcutaneous administration of 12600 ug of PDM608.
  6 subjects received PDM60.
- Part 1 SAD SC Placebo Cohort 5: One time subcutaneous administration of 12600 ug of PDM608.
  2 subjects received Placebo.
- Part 2 MAD SC PDM608 Cohort 1: Subcutaneous administration of 6300ug of PDM608/Placebo once weekly for 4 weeks.
  9 subjects received PDM608
- Part 2 MAD SC Placebo Cohort 1: Subcutaneous administration of 6300ug of PDM608/Placebo once weekly for 4 weeks.
  3 subjects received Placebo
- Part 2 MAD SC PDM608 Cohort 2: Subcutaneous administration of 12600ug of PDM608/Placebo once weekly for 4 weeks.
  9 subjects received PDM608 on week 1. 2 subjects were withdrawn per PI's discretion before receiving all 4 weekly doses of PDM608.
- Part 2 MAD SC Placebo Cohort 2: Subcutaneous administration of 12600ug of PDM608/Placebo once weekly for 4 weeks.
  3 subjects received Placeb
Period: Overall Study
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Started | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 9 | 3
Completed | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Two subjects from MAD Cohort 2 (both assigned to receive PDM608) did not complete the study and are excluded.
Groups:
- Part 1 SAD SC PDM608 Cohort 1: Single SC administration dose of 350 ug PDM608
- Part 1 SAD SC PDM608/Placebo Cohort 1: Single SC administration dose of 350 ug Placebo
- Part 1 SAD SC PDM608 Cohort 2: Single SC administration dose of 1050 ug PDM608
- Part 1 SAD SC Placebo Cohort 2: Single SC administration dose of 1050 ug Placebo
- Part 1 SAD SC PDM608Cohort 3: Single SC administration dose of 3150 ug PDM608
- Part 1 SAD SC Placebo Cohort 3: Single SC administration dose of 3150 ug Placebo
- Part 1 SAD SC PDM608 Cohort 4: Single SC administration dose of 6300 ug PDM608
- Part 1 SAD SC Placebo Cohort 4: Single SC administration dose of 6300 ug Placebo
- Part 1 SAD SC PDM608 Cohort 5: Single SC administration dose of 12600 ug PDM608
- Part 1 SAD SC Placebo Cohort 5: Single SC administration dose of 12600 ug Placebo
- Part 2 MAD SC PDM608 Cohort 1: Once a week subcutaneous administration of 6300 ug of PDM608 for 4 weeks
- Part 2 MAD SC Placebo Cohort 1: Once a week subcutaneous administration of 6300 ug of Placebo for 4 weeks
- Part 2 MAD SC PDM608 Cohort 2: Once a week subcutaneous administration of 12600 ug of PDM608 for 4 weeks
- Part 2 MAD SC Placebo Cohort 2: Once a week subcutaneous administration of 12600 ug of Placebo for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC PDM608/Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2 | Total
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3 | 62
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 15
  Male | 4 | 2 | 5 | 1 | 5 | 1 | 4 | 1 | 5 | 2 | 7 | 2 | 6 | 2 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3 | 62
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 9
  White | 5 | 2 | 6 | 2 | 5 | 2 | 4 | 1 | 4 | 2 | 8 | 3 | 7 | 2 | 53
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be analyzed for severity and potential relationship to PDM608 to determine safety and tolerability of PDM608
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Groups:
- Part 2 SAD SC Placebo Cohort 1: Single SC administration dose of 350 ug Placebo
- Part 1 SAD SC PDM608 Cohort 3: Single SC administration dose of 3150 ug PDM608
- Part 2 MAD SC PDM608 Cohort 2: Once a week subcutaneous administration of 12600 ug of PDM608 for 4 weeks
  2 subjects withdrew from the study prior to receiving all 4 weekly doses of PDM608.
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 2 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Test Results
Description: Results outside of laboratory defined normal ranges will be analyzed for clinical significance and used to determine safety and tolerability of PDM608
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 SAD SC Placebo Cohort 1: Single SC administration dose of 350 ug Placebo
- Part SAD SC Placebo Cohort 2: Single SC administration dose of 1050 ug Placebo
- Part SAD SC Placebo Cohort 3: Single SC administration dose of 3150 ug Placebo
- Part 1 SAD PDM608 Cohort 5: Single SC administration dose of 12600 ug PDM608
- Part 1 SAD Placebo Cohort 5: Single SC administration dose of 12600 ug Placebo
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD PDM608 Cohort 5 | Part 1 SAD Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Electrocardiogram Readings: QTcF
Description: Abnormal QTcF interval
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 SAD SC PDM608 Cohort 2; Part 1 SAD SC Placebo Cohort 2: Single SC administration dose of 1050 ug Placebo
- Part 2 MAD SC PDM608 Placebo Cohort 2: Once a week subcutaneous administration of 12600 ug of Placebo for 4 weeks
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC PDM608 Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Electrocardiogram Readings: VR
Description: Abnormal ventricular rate
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 SAD SC PDM608Cohort 5: Single SC administration dose of 12600 ug PDM608
- Part 2 MAD SC PDM608 Cohort 1: Multiple ascending dose, subcutaneous once weekly for 4 weeks administration of 6300 ug PDM608
- Part 2 MAD SC Placebo Cohort 1: Multiple ascending dose, subcutaneous once weekly for 4 weeks administration of 6300 ug Placebo
- Part 2 MAD SC Placebo Cohort 2: Once a week subcutaneous administration of 12600 ug of PDM608/Placebo for 4 weeks
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Electrocardiogram Readings: PR Interval
Description: Abnormal PR interval
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Electrocardiogram Readings: QRS Duration
Description: Abnormal QRS duration
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Electrocardiogram Readings: QRS Axis
Description: Abnormal QRS axis
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Abnormal Vital Signs: BP
Description: Abnormal systolic and/or diastolic pressure (mmHg)
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Abnormal Vital Signs: HR
Description: Abnormal heart rate (beats/minute)
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 SAD Placebo Cohort 3: Single SC administration dose of 3150 ug Placebo
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Abnormal Vital Signs: Temp
Description: Abnormal body temperature (Celsius)
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 SAD SC Placebo Cohort 3: Single SC administration dose of 3150 ug Placebos
- Part 1 SAD SC Placebo Cohort 4: Single SC administration dose of 6300 ug PDM608
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Abnormal Vital Signs: RR
Description: Abnormal respiratory rate (breaths/minute)
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Abnormal Physical Exams
Description: Physical exams will include evaluation of general appearance, head, neck, thyroid, eyes, ears, nose and throat, respiratory, cardiovascular, abdomen, dermatological, genitourinary, musculoskeletal and neurological systems
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 9 | 3 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Assess PK Parameters for Single (Part 1) and Multiple (Part 2) SC Doses of PDM608 in Healthy Volunteers.
Description: Analysis of PDM608 plasma concentration data will be performed using PK parameters.
Time Frame: Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26
Population: Cmax for subjects dosed with PDM608
  Following a single SC administration of PDM608 at dose levels of 350 μg (cohort 1) and 1050 μg (cohort 2), serum concentrations of PDM608 were BLQ (<10.0 ng/mL) for all subjects and time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 1 SAD SC PDM608 Cohort 1: Single SC administration dose of 350 ug PDM608/Placebo
- Part 1 SAD SC PDM608 Cohort 2: Single SC administration dose of 1050 ug PDM608/Placebo
- Part 1 SAD SC PDM608 Cohort 3: Single ascending dose, subcutaneous administration of PDM608 dose of 3150 ug
- Part 1 SAD SC PDM608 Cohort 4: Single ascending dose, subcutaneous administration of PDM608 dose of 6300 ug
- Part 1 SAD SC PDM608 Cohort 5: Single ascending dose, subcutaneous administration of PDM608 dose of 12600 ug
- Part 2 MAD SC PDM608 Cohort 1 Day 1: Subcutaneous dose of 6300 ug PDM608/Placebo-post first weekly dose.
- Part 2 MAD SC PDM608 Cohort 1 Day 22: Subcutaneous dose of 6300 ug PDM608/Placebo-post 4th and final weekly dose.
- Part 2 MAD SC PDM608 Cohort 2 Day 1: Subcutaneous dose of 12600 ug PDM608/Placebo-post first weekly dose.
- Part 2 MAD S CPDM608 Cohort 2 Day 22: Subcutaneous dose of 12600 ug PDM608/Placebo-post fourth and final weekly dose.
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 Day 1 | Part 2 MAD SC PDM608 Cohort 1 Day 22 | Part 2 MAD SC PDM608 Cohort 2 Day 1 | Part 2 MAD S CPDM608 Cohort 2 Day 22
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 8
ng/mL | NA (NA) — below the level of detection | NA (NA) — below the level of detection | 23.4 (52.2) | 52.4 (96.4) | 203 (70.5) | 44.2 (60.2) | 21.9 (247.9) | 150 (0) | 10.7 (0)

14. Secondary Outcome: To Assess Immunogenicity Following Single and Multiple Doses of PDM608
Description: Incidence of ADA in blood
Time Frame: Part 1: Day 1 through Day 22; Part 2: Day 1 through Day 60
Population: The Number of Participants with Positive Anti-Drug Antibodies. Data was not collected for SAD cohorts for 144 and 912 hours pose dose. Data was not collected for MAD cohorts 1-2 for 336 and 504 hours post dose.
Measure: Number; unit: participants
Groups:
- Part 1 SAD SC PDM608 Cohort 1: Single ascending dose, subcutaneous administration of 350 ug PDM60 dose
- Part 1 SAD SC PDM608 Cohort 2: Single ascending dose, subcutaneous administration of 1050 ug PDM608
- Part 1 SAD SC PDM608 Cohort 3: Single ascending dose, subcutaneous administration of 3150 ug PDM608
- Part 1 SC PDM608 Cohort 4: Single ascending dose, subcutaneous administration of 6300 ug PDM608
- Part 1 SAD SC PDM608 Cohort 5: Single ascending dose, subcutaneous administration of 12600 ug PDM608
- Part 2 MAD SC PDM608 Cohort 1: Multiple ascending dose, subcutaneous once weekly for 4 weeks administration of 6300 ug PDM608.
  Cohort 2: 12600 ug.
- Part 2 MAD SC PDM608 Cohort 2: Multiple ascending dose, subcutaneous once weekly for 4 weeks administration of 12600 ug PDM608.
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SC PDM608 Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC PDM608 Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 9 | 9
participants
  336 hours post-dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0 | 0
  336 hours post-dose | 4 | 6 | 5 | 5 | 6 |  |
  504 hours post-dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0 | 0
  504 hours post-dose | 4 | 5 | 5 | 6 | 6 |  |
  Day 28 (144 hours post-dose): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 9
  Day 28 (144 hours post-dose) |  |  |  |  |  | 9 | 7
  Day 60 (912 hours post-dose): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 9
  Day 60 (912 hours post-dose) |  |  |  |  |  | 7 | 7

ADVERSE EVENTS:
Time Frame: Adverse events was collected from the time of consent to 30 days after the last dose of study drug. For Part 1, duration of study participation is 22 days with PDM608/Placebo administered on Day 1. Study duration for Part 2 is 60 with the last dose of PDM608/Placebo administered on Day 22. If subjects have ongoing AEs at the end of study visit, the study team contacted the subjects weekly until AE resolution.
Description: During each study visit, subjects were questioned directly regarding occurrence of any adverse medical event. All AEs were documented in the EDC, including date, time of onset, description of AE, severity, seriousness, duration, actions taken, outcome and an investigator's opinion on relationship between study drug.
Arm/Group | Part 1 SAD SC PDM608 Cohort 1 | Part 1 SAD SC Placebo Cohort 1 | Part 1 SAD SC PDM608 Cohort 2 | Part 1 SAD SC Placebo Cohort 2 | Part 1 SAD SC PDM608 Cohort 3 | Part 1 SAD SC Placebo Cohort 3 | Part 1 SAD SC PDM608 Cohort 4 | Part 1 SAD SC Placebo Cohort 4 | Part 1 SAD SC PDM608 Cohort 5 | Part 1 SAD SC Placebo Cohort 5 | Part 2 MAD SC PDM608 Cohort 1 | Part 2 MAD SC Placebo Cohort 1 | Part 2 MAD SC PDM608 Cohort 2 | Part 2 MAD SC Placebo Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/9 | 0/3 | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/9 | 0/3 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 5/6 | 0/2 | 5/6 | 1/2 | 4/6 | 0/2 | 6/6 | 0/2 | 6/6 | 0/2 | 9/9 | 2/3 | 9/9 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 SAD SC PDM608 Cohort 1 (N=6) | Part 1 SAD SC Placebo Cohort 1 (N=2) | Part 1 SAD SC PDM608 Cohort 2 (N=6) | Part 1 SAD SC Placebo Cohort 2 (N=2) | Part 1 SAD SC PDM608 Cohort 3 (N=6) | Part 1 SAD SC Placebo Cohort 3 (N=2) | Part 1 SAD SC PDM608 Cohort 4 (N=6) | Part 1 SAD SC Placebo Cohort 4 (N=2) | Part 1 SAD SC PDM608 Cohort 5 (N=6) | Part 1 SAD SC Placebo Cohort 5 (N=2) | Part 2 MAD SC PDM608 Cohort 1 (N=9) | Part 2 MAD SC Placebo Cohort 1 (N=3) | Part 2 MAD SC PDM608 Cohort 2 (N=9) | Part 2 MAD SC Placebo Cohort 2 (N=3)
Injection Site Reactions (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 5 (9) | 1 (1) | 4 (8) | 0 (0) | 6 (10) | 0 (0) | 6 (8) | 0 (0) | 9 (34) | 2 (3) | 9 (35) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT05950906/Prot_SAP_000.pdf